CLINICAL TRIAL: NCT05340075
Title: Staged Bilateral Percutaneous Nephrolithotomy: When to Operate for a Contralateral Kidney?
Brief Title: Staged Bilateral Percutaneous Nephrolithotomy
Status: Completed | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ali Kaan Yildiz, Principal Investigator, Ankara Training and Research Hospital
Other Study IDs: PCNL2022
Record Dates: First submitted 2022-03-30; First posted 2022-04-21 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Stone, Kidney; Urolithiasis
MeSH Terms: conditions — Kidney Calculi; Urolithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Staged percutaneous nephrolithotomy group 1: Those who underwent percutaneous nephrolithotomy 2-4 weeks after percutaneous nephrolithotomy for stones in the other kidney
  Interventions: Procedure: Patients who underwent percutaneous nephrolithotomy
- Staged percutaneous nephrolithotomy group 2: Those who underwent percutaneous nephrolithotomy 4-6 weeks after percutaneous nephrolithotomy for stones in the other kidney
  Interventions: Procedure: Patients who underwent percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: Patients who underwent percutaneous nephrolithotomy — Patients who underwent percutaneous nephrolithotomy to the contralateral kidney 2-4 weeks and 4-6 weeks after the percutaneous nephrolithotomy operation

SUMMARY:
To determine the optimal time between the first and second operations in patients with bilateral kidney stones and scheduled percutaneous nephrolithotomy for the contralateral kidney. Patients who underwent percutaneous nephrolithotomy to the contralateral kidney 2-4 weeks and 4-6 weeks after the first operation will be compared.

DETAILED DESCRIPTION:
The aim of the study is to determine the optimal time between the first and second operations in patients with bilateral kidney stones and scheduled percutaneous nephrolithotomy for the contralateral kidney. In our study, patients who underwent percutaneous nephrolithotomy to the contralateral kidney 2-4 weeks and 4-6 weeks after the first operation will be compared. With the guidance of preoperative and postoperative data, it is aimed to determine the optimal time with the lowest complication and highest operational success.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stones of 2 cm or more in each kidney

Exclusion Criteria:

* Renal Failure
* Coagulopathy
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stones of 2 cm or more in each kidney
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
BMI in kg/m^2 | 3 Months
  BMI in kg/m^2
rates of intraoperative blood transfusion, operation time(minute) | 3 Months
  rates of intraoperative blood transfusion, operation time(minute)

SECONDARY OUTCOMES:
mm size of the stone, | 3 Months
  mm size of the stone,

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wollin DA, Preminger GM. Percutaneous nephrolithotomy: complications and how to deal with them. Urolithiasis. 2018 Feb;46(1):87-97. doi: 10.1007/s00240-017-1022-x. Epub 2017 Nov 17. PMID 29149365
- [Background] ElSheemy MS, Ghoneima W, Elmarakbi AA, Al-Kandari AM, Ibrahim H, Shrestha S, Khadgi S. Bilateral Single-session vs Staged Mini-percutaneous Nephrolithotomy for Renal Stones: A Comparative Study. Urology. 2018 Oct;120:62-67. doi: 10.1016/j.urology.2018.07.015. Epub 2018 Jul 20. PMID 30031834
- [Background] Torricelli FCM, Carvalho RS, Marchini GS, Danilovic A, Vicentini FC, Batagello CA, Srougi M, Nahas WC, Mazzucchi E. Bilateral simultaneous percutaneous nephrolithotomy versus staged approach: a critical analysis of complications and renal function. Rev Assoc Med Bras (1992). 2020 Dec;66(12):1696-1701. doi: 10.1590/1806-9282.66.12.1696. PMID 33331579